CLINICAL TRIAL: NCT04890808
Title: Therapeutic Antioxidant Supplementation for Enhancement of Neural Protection From Free-iron Toxicity in Superficial Siderosis
Brief Title: Therapeutic Antioxidant Supplementation
Acronym: TAS-SS21
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superficial Siderosis Research Alliance Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SSRA0921
Record Dates: First submitted 2021-05-12; First posted 2021-05-18 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2021-05

CONDITIONS: Superficial Siderosis
Keywords: Hemosiderin; Iron Toxicity; Superficial siderosis of the CNS; Infratentorial superficial siderosis; Neurodegenerative disorder; Subpial
MeSH Terms: conditions — Neurodegenerative Diseases | interventions — Inosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Over-the-Counter Dietary Supplement Inosine (Experimental): capsules containing 500 mg of inosine Two capsules Twice Daily Other Name: hypoxanthine 9-β-D-ribofuranoside 9-[(2R,3R,4S,5R)-3,4-dihydroxy-5-hydroxymethyl) oxolan-2-yl]-1H-purin-6-one
  Interventions: Dietary Supplement: Inosine
- Over-the-Counter Dietary Supplement IP6 (Experimental): capsules containing 500mg of IP6 Two capsules Twice Daily Other Name: Inositol hexaphosphate
  (1R,2S,3r,4R,5S,6s)-cyclohexane-1,2,3,4,5,6-hexayl hexakis[dihydrogen (phosphate)]
  Interventions: Dietary Supplement: IP6

INTERVENTIONS:
Dietary Supplement: Inosine — Patients will be dosed with two 500 mg capsules of Inosine twice daily for 36 months
  Arms: Over-the-Counter Dietary Supplement Inosine
Dietary Supplement: IP6 — Patients will be dosed with two 500 mg capsules of IP6 twice daily for 36 months
  Arms: Over-the-Counter Dietary Supplement IP6

SUMMARY:
A remotely administered study, non-randomized, non-blinded, controlled parallel assignment phase 2 trial to determine if oral inosine or inositol hexaphosphate will provide an effective long-term therapy to combat or slow neural damage progression either concurrently with existing iron chelation therapy or during the natural course of the disorder. Clinical changes in hearing, balance, and mobility, and cognition will be assessed for 36 months through patient-reported outcomes of study assigned assessments.

DETAILED DESCRIPTION:
Capsules containing over-the-counter dietary supplement formulas of inosine 500 mg or 500 mg of inositol hexaphosphate(IP6) will be taken orally, two capsules two times per day for 36 months. Initial screening will determine patient arm assignment.

Before dosing begins, patients will submit copies of previous audiogram results (3yrs), radiology reports (3yrs), and MRI series (3yrs) if available and complete baseline assessment activities: Montreal Cognitive Assessment (MoCA) administered remotely, Timed Up, and Go (TUG), 2-Minute Walk Test (2-MWT), The Activities-specific Balance Confidence (ABC) Scale, iSS-QoL (custom) patient outcome reported

Assessment will take place four times: baseline, end-of-year 1 (12mo), end-of-year 2 (24mo), end-of-study (36mo).

ELIGIBILITY:
Inclusion Criteria:

Confirmed diagnosis of iSS (superficial siderosis of the CNS)

No illegal drug use

No history of myocardial infarction or stroke

No history of severe chronic obstructive pulmonary disease

Can safely swallow large capsules

Exhibits at least one confirmed iSS related symptom: Hearing Loss, Balance, Memory/Cognitive problems

Does not have a known hypersensitivity or intolerance to any study antioxidant

Has not taken part in another treatment study for any condition within the last 30 days (about four and a half weeks)

Not currently pregnant or breastfeeding

Exclusion Criteria:

Inosine Arm Exclusion :

Diagnosed with urate urolithiasis, or recurrent urolithiasis, all unknown type

History of Gout

History of Kidney Stones

P6 Arm Exclusion

Long-term anticoagulant

Known or suspected active bleed into the CNS

Currently undergoing deferiprone chelation therapy

Plan to begin deferiprone chelation therapy within three years

-

Ages: 16 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Slow the Rate of Clinical Decline | 36 Months
  Deceleration of clinical decline will be quantified by evaluating three primary areas- hearing, balance and mobility, and cognition. End-of-study quantifiable slowing of the historical and year-1 mean rate of decline across all three study areas with a measurable increase on Year-3 iSS-QOL from Year-1 iSS-QOL scoring.

SECONDARY OUTCOMES:
Clinical Efficacy: Rate of Adverse Event Development [Safety and Tolerability} | 36 Months
  Therapeutic use of antioxidants through a safe, effective dose range and schedule to the extent that the risk-benefit relationship is acceptable for the patient. Evaluation will include the overall adverse event (AE) and serious AE (SAE) rate.
Clinical Efficacy: Improved Quality of Life | 36 Months
  The rate of change in points on the iSS-QoL(custom) from baseline assessment to end-of-study will be scored based on 16 questions with a point range of 1-5. Higher end-of-study scores indicate greater satisfaction.
Clinical Efficacy: Rate of Change in Montreal Cognitive Assessment (MoCA) | 36 Months
  The rate of change in points on the Montreal Cognitive Assessment (MoCA) scale from baseline assessment to end-of-study will be assessed for patients in each treatment group. The MoCA assesses attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Points (range 0-30) are awarded for the correct completion of MoCA tasks. Cognition decline will be defined as ≥ 3pt decline of total MoCA score from baseline assessment to final 36mo testing assessment.
Clinical Efficacy: Rate of Change in Hearing | 36 Months
  The baseline audiogram will be compared to the post-study audiogram for each patient. The hearing levels in decibels against the frequency in hertz will be compared pre-study, baseline, and end-of-study for average rate-of-decline. A paired t-test will be used to determine statistical significance in the average difference in the threshold hearing level at any particular frequency.
Clinical Efficacy: Rate of Change in Mobility and Balance | 36 Months
  The Timed Up & Go (TUG), 2-Minute Walk Test (2MWT), and Activities-specific Balance Confidence (ABC) Scale will be scored individually. The baseline score will be compared to the annual and end-of-study scores for each patient. A paired t-test will be used to determine statistical significance in the average difference.
Clinical Efficacy: Hemosiderin Reduction (IP6 Arm) | 36 Months
  Visible hemosiderin deposition reduction on MRI series from baseline visit to end-of-study. MRIs will be objectively analyzed for changes in iron deposition.

CONTACTS AND LOCATIONS:
Overall Officials: Rori-Suzanne Daniel, Study Director — Superfical Siderosis Research Alliance

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Superficial Siderosis Patient Registry — https://superficialsiderosis.org
- See also: Superficial Siderosis research Alliance — https://ssra.livingwithss.com